CLINICAL TRIAL: NCT01793181
Title: Vitamin D Levels in Patients With Central Retinal Vein Occlusion- a Prospective Controlled Study
Status: Completed | Type: Observational
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Anders Kvanta, Associate Professor, St. Erik Eye Hospital
Other Study IDs: 201149311
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Vitamin d Deficiency; Central Retinal Vein Occlusion
Keywords: Vitamin d deficiency; Central retinal vein occlusion
MeSH Terms: conditions — Vitamin D Deficiency; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample of vitamin D
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CRVO patients: Patients with a newly diagnosed CRVO. Maximum duration 3 months.
- Control patients: Controls matched for age,gender, month of onset from the Central Bureau of Statistics Sweden

SUMMARY:
Retinal vein occlusion (RVO) is a common vascular disease of the eye. Studies have shown that the risk of venous thrombosis is higher in winter so even concerning RVO. Studies have shown a possible link between sun exposure and venous thrombosis. Vitamin D levels have been shown to have a similar seasonal variation, with a peak occurring in the summer. The primary source of vitamin D is from sunlight when ultraviolet B (UVB) radiation penetrates the skin and converts 7-dehydrocholesterol to 25-hydroxycholecalciferol vitamin D3 (25-OHVitD) via previtamin D. In Stockholm situated at latitude 59˚ 20΄ North, it is not possible to synthesize vitamin D at sufficient levels in winter and the exposure time required to reach a standard dose is impractical from at least October through March.

The aim of the study is to evaluate vitamin D levels in central retinal vein occlusion (CRVO) patients and compare them with the vitamin D levels in randomly selected control patients matched for age and month of disease onset. This is to evaluate whether vitamin D deficiency may be a risk factor in the onset of CRVO.

The hypothesis of the study is that patients with CRVO have lower levels of vitamin d than matched controls.

DETAILED DESCRIPTION:
The study will last one year and is expected to include 120 patients with RVO and 120 control patients. The first 10 RVO patients visiting St. Erik's Eye Hospital with disease duration of maximum 3 months will be included in the study each month. The control patients will be chosen randomly by the Central Bureau of Statistics and matched for age and gender according to disease distribution known from previous studies. The control group will receive a letter with information of the study, informed consent form and details about the blood sampling procedure. Every month 50 patients in the control group will be invited to participate in the study. Only the first 10 control subjects will be included in the study. Each month a blood sample will be taken from 10 patients with RVO and 10 subjects in the control group. All the subjects will only have one blood sample taken during the study. Blood will be analyzed to measure the vitamin D level. Vitamin D levels will be compared at the end of the study between groups and evaluated according to the time of year for sampling. All the blood sampling will be done by the laboratory at Karolinska University Hospital. Participation in the study is completely voluntary. The details of the study has been reviewed and approved by the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed central retinal vein occlusion (3 months)

Exclusion Criteria:

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with central retinal vein occlusion diagnosed at St Eriks Eye Hospital
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels | one year

CONTACTS AND LOCATIONS:
Locations (1):
- St Eriks Eye Hospital, Stockholm, Stockholm County, Sweden